CLINICAL TRIAL: NCT03687281
Title: Pilot Study on Practice of "Chemical Sex" by Men Having Sex With Men Living With HIV Followed at Reunion Island University Hospital Center
Brief Title: Practice of "Chemical Sex" by HIV Patients in Reunion Island
Acronym: CHEMSEX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/CHU/03
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: HIV
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients living with HIV and having sex with men: Male patients living with HIV and having sex with men followed at Universitary Hospital Center of Reunion Island
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The questionnaire consists of three parts:
  * knowledge assessment;
  * socio-demographic, medical and lifestyle data;
  * use of "Chemsex".
  Other Names: CHEMSEX questionnaire

SUMMARY:
The term "CHEMSEX", short for "chemicals" and "sex", is used to define the consumption, regardless of the route of administration, of drugs or substances for recreational use, in a sexual context.

No published data is currently available concerning this practice in Reunion Island. However, an upsurge in cases of acute hepatitis C was observed at the end of 2016 (4 in 6 months) of which 3 were related to the practice of chemsex (data CeGGID Réunion) and the recent years have been marked by many cases related to drug trafficking and the arrival of substances still unknown on the island.

Given the rapid emergence of the phenomenon in metropolitan France and in the rest of the world, serious consequences that are both psychological, addictological and infectious, to take stock of this practice among MSM patients followed in Reunion Island seems essential. to establish a rapid, adequate and effective prevention and action plan.

DETAILED DESCRIPTION:
The term "CHEMSEX", short for "chemicals" and "sex", is used to define the consumption, regardless of the route of administration, of drugs or substances for recreational use, in a sexual context.

Although the use of drugs and narcotics is not a novelty in sexual practice, however, there is a change in behavior. Indeed, the advent of synthetic products such as cathinones, easily obtained via the internet and at affordable prices has attracted a wider audience and has allowed in less than ten years, the amplification of this worrying phenomenon.

The described effects of cathinones are just as powerful as the classic drugs that were quickly supplanted: intellectual stimulation, exacerbation of the senses, euphoria, disinhibition, sexual arousal, relaxation.

These initially ingested or inhaled products are quickly injected for a greater rapidity of their hallucinogenic and psychostimulant effects. SLAM ("slap"), is the Anglo-Saxon term commonly used to describe the intravenous use of drugs in the context of sexual practices. The subjects are gradually led to modify and increase their consumption, for ever more effect.

The consequences of this practice are multiple and serious: addiction with all the risks incurred, psychiatric and infectious complications related to the sharing of contaminated material (endocarditis, hepatitis ...) and unprotected sex ratios favoring the transmission of STIs.

In the literature, all the studies on the subject concern men having sex with men, and more particularly patients living with HIV. Indeed, the prevalence of HIV is 70 to 82% among these practitioners.

European studies, particularly in London gay festive environnement, show the increasing use of these substances resulting in risky behavior. In recent years, STIs have been increasing and more particularly in the men having sex with men population.

No published data is currently available concerning this practice in Reunion Island. However, an upsurge in cases of acute hepatitis C was observed at the end of 2016 (4 in 6 months) of which 3 were related to the practice of chemsex (data CeGGID Réunion) and the recent years have been marked by many cases related to drug trafficking and the arrival of substances still unknown on the island.

Given the rapid emergence of the phenomenon in metropolitan France and in the rest of the world, serious consequences that are both psychological, addictological and infectious, to take stock of this practice among MSM patients followed in Reunion Island seems essential. to establish a rapid, adequate and effective prevention and action plan.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Man having sex with men;
* Patients living with HIV;
* Followed at Universitary Hospital Center of Reunion Island;
* Able to answer a self-questionnaire in French;
* Having agreed to participate

Exclusion Criteria:

* Subject under legal protection;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients living with HIV and having sex with men
Study Population: Patients living with HIV followed in Clinical Immunology service of Universitary Hospital Centre in Reunion Island
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of recent chemsex practice | Day 1
  Proportion of subjects practicing chemsex on and off department (practice over the last 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion